CLINICAL TRIAL: NCT01212757
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Efficacy and Safety Study of Two Doses of Apremilast (CC-10004) in Subjects With Active Psoriatic Arthritis
Brief Title: PALACE 2: Efficacy and Safety Study of Apremilast to Treat Active Psoriatic Arthritis
Acronym: PALACE2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSA-003; 2010-018386-32 (EudraCT Number)
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriasis; Arthritis; Psoriatic Arthritis; inflammation; skin condition; inflammatory cells; apremilast; CC-10004; phosphodiesterase type 4
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Arthritis; Inflammation; Skin Diseases | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Apremilast 20mg (Experimental): 20 mg Apremilast tablets administered twice daily for 24 weeks during the placebo-controlled phase followed by 20 mg Apremilast tablets administered twice daily for up to 4.5 years in the active treatment / long-term safety phase
  Interventions: Drug: Apremilast 20mg
- Apremilast 30mg (Experimental): 30 mg Apremilast tablets administered twice a day for 24 weeks during the placebo-controlled phase followed by 30 mg Apremilast tablets administered twice a day for up to 4.5 years in the active treatment / long-term safety phase orally twice daily
  Interventions: Drug: Apremilast 30mg
- Placebo + 20 mg Apremilast (Placebo Comparator): Placebo + 20 mg Apremilast tablets administered twice daily for 24 weeks during the placebo-controlled phase followed by 20 mg Apremilast tablets administered twice daily for up to 4.5 years in the active treatment / long-term safety phase. Subjects who do not have at least 20% improvement in their swollen and tender joint counts at Week 16 will escape to 20 mg Apremilast twice daily at Week 16
  Interventions: Drug: Placebo + 20 mg Apremilast
- Placebo + 30 mg Apremilast (Placebo Comparator): Placebo + 30 mg Apremilast tablets administered twice daily for 24 weeks during the placebo-controlled phase followed by 30 mg Apremilast tablets administered twice daily for up to 4.5 years in the active treatment / long-term safety phase. Subjects who do not have at least 20% improvement in their swollen and tender joint counts at Week 16 will escape to 30 mg Apremilast twice daily at Week 16.
  Interventions: Drug: Placebo + 30 mg Apremilast

INTERVENTIONS:
Drug: Apremilast 20mg — Apremilast 20 mg twice daily, orally
  Other Names: CC-10004
  Arms: Apremilast 20mg
Drug: Apremilast 30mg — Apremilast 30 mg twice daily, orally
  Other Names: CC-10004
  Arms: Apremilast 30mg
Drug: Placebo + 20 mg Apremilast — Placebo + 20 mg Apremilast
  Other Names: Placebo; CC-10004
  Arms: Placebo + 20 mg Apremilast
Drug: Placebo + 30 mg Apremilast — Placebo + 30 mg Apremilast
  Other Names: Placebo; CC-10004
  Arms: Placebo + 30 mg Apremilast

SUMMARY:
The purpose of this study is to determine whether apremilast is safe and effective in the treatment of patients with psoriatic arthritis.

Apremilast is proposed to improve signs and symptoms of psoriatic arthritis (tender and swollen joints, pain, physical function) in treated patients.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is an inflammatory arthritis that occurs in 6-39% of psoriasis patients. The immunopathogenesis of PsA, which mirrors but is not identical to that seen in psoriatic plaques, reflects a complex interaction among resident dendritic, fibroblastic and endothelial cells, and inflammatory cells attracted to the synovium by cytokines and chemokines. Apremilast (CC-10004) is a novel oral agent that modulates multiple inflammatory pathways through targeted phosphodiesterase type 4 (PDE4) enzyme inhibition. Therefore, apremilast has the potential to be effective in the treatment of PsA.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged ≥ 18 years at time of consent.
* Have a diagnosis of Psoriatic Arthritis (PsA, by any criteria) of ≥ 6 months duration.
* Meet the Classification Criteria for Psoriatic Arthritis (CASPAR) PsA at time of screening.
* Must have been inadequately treated by disease-modifying antirheumatic drugs (DMARDs)
* May not have axial involvement alone
* Concurrent Treatment allowed with methotrexate, leflunomide, or sulfasalazine
* Have ≥ 3 swollen AND ≥ 3 tender joints.
* Males & Females must use contraception
* Stable dose of nonsteroidal anti-inflammatory drugs (NSAIDs), narcotics and low dose oral corticosteroids allowed.

Exclusion Criteria:

* Pregnant or breast feeding.
* History of allergy to any component of the investigational product.
* Hepatitis B surface antigen and/or Hepatitis C antibody positive at screening.
* Therapeutic failure on > 3 agents for PsA or > 1 biologic tumor necrosis factor (TNF) blocker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2010-09-27 (Actual); Primary Completion 2012-07-26 (Actual); Study Completion 2017-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (98):
- United States (23):
  - Clinical and Translational Research Center of Alabama, PC, Tuscaloosa, Alabama
  - Denver Arthritis Clinic, Denver, Colorado
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Centre For Rheumatology, Immun. And Arthritis, Fort Lauderdale, Florida
  - DMI Research, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Arthritis and Rheumatology of Georgia, Atlanta, Georgia
  - Michael Bukhalo MD SC, Arlington Hts, Illinois
  - Associated Internal Medical Specialist, PC, Battle Creek, Michigan
  - Advanced Rheumatology, Lansing, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Research West Incorporated, Kalispell, Montana
  - University of Rochester Medical Center, Rochester, New York
  - Vital Research, Greensboro, North Carolina
  - Unifour Medical Research Associatets LLC, Hickory, North Carolina
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas
  - Baylor Research Institute, Dallas, Texas
  - Arthritis Care and Diagnostic Center, Dallas, Texas
  - Luckster Enterprises, San Antonio, Texas
  - Seattle Rheumatology Associates, Seattle, Washington
  - Tacoma Center for Arthritis Research, PS, Tacoma, Washington
  - Rheumatology and Immunotherapy Center, Franklin, Wisconsin
- Belgium (4):
  - CHU Brugmann, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - University Hospital of Liege CHU Liege, Liège
- Bulgaria (6):
  - Diagnostic and Consulting Centre 7, Sofia
  - University Multiprofile Hospital for Active Treatment ACIBADEM City Clinic Sofia, Sofia
  - 17 Diagnostic and Consulting Centre Sofia EOOD, Sofia
  - Multiprofile Hospital for Active Treatment Sv. Ivan Rilski, Sofia
  - Diagnostic-Consultative Center Sveta Anna, Sofia
  - Diagnostic and Consulting Centre 4, Varna
- Canada (8):
  - Rheumatology Research Associates, Edmonton, Alberta
  - PerCuro Clinical Research, Victoria, British Columbia
  - Anna Jaroszynska Private Practice, Burlington, Ontario
  - William Bensen's Private Practice, Hamilton, Ontario
  - North Bay Dermatology Center, North Bay, Ontario
  - Rheumatology Research Associates, Ottawa, Ontario
  - Wilderman Medical Clinic, Thornhill, Ontario
  - Darryl Toth's Private Practice, Windsor, Ontario
- Czechia (9):
  - Revmatologie s.r.o., Brno
  - MEDIPONT PLUS s.r.o.., České Budějovice
  - L.K.N. Arthrocentrum s.r.o., Hlučín
  - ARTMEDI UPD s.r.o., Hostivice
  - Revmatologicky ustav, Prague
  - Revmatologicka Ambulance, Prague
  - Affidea Praha s.r.o, Prague
  - Revmatologicka Ambulance, Sokolov
  - PV - MEDICAL, s.r.o., Zlín
- Estonia (5):
  - Parnu Hospital, Pärnu
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Regional Hospital, Tallinn
  - Clinical Research Centre Ltd, Tartu
  - Tartu University Hospital, Tartu
- France (5):
  - Hopital Universitaire Dupuytren, Limoges
  - Hopital Lariboisiere, Paris
  - Fondation Hôpital Saint-Joseph, Paris
  - Groupe Hospitalier Pitié- Salpétrière, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (4):
  - Charite - Universitätsmedizin Berlin, Berlin
  - Klinikum der Johann-Wolfgang Goethe-Universität, Frankfurt
  - Praxis Karin Rockwitz, Goslar
  - Synexus Clinical Research GmbH, Leipzig
- Hungary (3):
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Principal SMO Kft., Makó
- Italy (6):
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Ospedale Luigi Sacco, Milan
  - Seconda Universita degli Studi di Napoli, Napoli
  - IRCCS Policlinico San Matteo, Pavia
  - Universita di Pisa, Pisa
  - Ospedale Civile Maggiore Borgo Trento, Verona
- Poland (5):
  - NZOZ Osteo-Medic sc A. Racewicz J. Supronik, Bialystok
  - Niepubliczny Zaklad Opieki Zdrowotnej REUMED, Lublin
  - Wojskowy Instytut Medyczny, Warsaw
  - Instytut Reumatologii im. prof. dr hab. med. Eleonory Reicher, Warsaw
  - Synexus SCM Sp. z o.o., Wroclaw
- Russia (4):
  - City Clinical Hospital #1 n.a. N.I.Pirogov, Moscow
  - City Clinical Hospital #5, Nizhny Novgorod
  - St.Petersburg State Medical Academy n. a. I.I.Mechnikov, Saint Petersburg
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
- South Africa (3):
  - Nelson Mandela School Of Medicine, Durban
  - Greenacres Hospital, Port Elizabeth
  - Jacaranda Hospital, Pretoria
- Spain (3):
  - Hospital General Carlos Haya, Málaga
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Sierrallana, Torrelavega
- Taiwan (5):
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Cathay General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Tapei
- United Kingdom (5):
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Cannock Chase Hospital, Cannock
  - Chapel Allerton Hospital, Leeds
  - Poole Hospital, Poole
  - Great Western Hospital, Swindon

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Cutolo M, Myerson GE, Fleischmann RM, Liote F, Diaz-Gonzalez F, Van den Bosch F, Marzo-Ortega H, Feist E, Shah K, Hu C, Stevens RM, Poder A. A Phase III, Randomized, Controlled Trial of Apremilast in Patients with Psoriatic Arthritis: Results of the PALACE 2 Trial. J Rheumatol. 2016 Sep;43(9):1724-34. doi: 10.3899/jrheum.151376. Epub 2016 Jul 15. PMID 27422893
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690
- [Derived] Mease PJ, Gladman DD, Kavanaugh A, McGonagle D, Nash P, Guerette B, Nakasato P, Brunori M, Teng L, McInnes IB. Articular and Extra-Articular Benefits in ACR20 Non-responders at Week 104 Treated With Apremilast: Pooled Analysis of Three Randomized Controlled Trials. Rheumatol Ther. 2021 Dec;8(4):1677-1691. doi: 10.1007/s40744-021-00369-x. Epub 2021 Sep 18. PMID 34536218
- [Derived] Mease PJ, Gladman DD, Ogdie A, Coates LC, Behrens F, Kavanaugh A, McInnes I, Queiro R, Guerette B, Brunori M, Teng L, Smolen JS. Treatment-to-Target With Apremilast in Psoriatic Arthritis: The Probability of Achieving Targets and Comprehensive Control of Disease Manifestations. Arthritis Care Res (Hoboken). 2020 Jun;72(6):814-821. doi: 10.1002/acr.24134. Epub 2020 May 8. PMID 31909868
- [Derived] Kavanaugh A, Gladman DD, Edwards CJ, Schett G, Guerette B, Delev N, Teng L, Paris M, Mease PJ. Long-term experience with apremilast in patients with psoriatic arthritis: 5-year results from a PALACE 1-3 pooled analysis. Arthritis Res Ther. 2019 May 10;21(1):118. doi: 10.1186/s13075-019-1901-3. PMID 31077258
- [Derived] Gladman DD, Kavanaugh A, Gomez-Reino JJ, Wollenhaupt J, Cutolo M, Schett G, Lespessailles E, Guerette B, Delev N, Teng L, Edwards CJ, Birbara CA, Mease PJ. Therapeutic benefit of apremilast on enthesitis and dactylitis in patients with psoriatic arthritis: a pooled analysis of the PALACE 1-3 studies. RMD Open. 2018 Jun 27;4(1):e000669. doi: 10.1136/rmdopen-2018-000669. eCollection 2018. PMID 30018799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a multicenter study with 84 sites from the United States, Canada, Europe, Russia, Australia, South Africa and Taiwan.
Pre-assignment Details: This study consisted of a 24-week randomized, double-blind, placebo-controlled phase, a 28-week randomized, double-blind active treatment phase and a 4-year open-label safety phase, for an overall study duration of 5 years.
Groups:
- Placebo: Participants initially randomized to placebo tablets twice daily (BID) in the 24-week placebo-controlled phase. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were re-randomized to either 20 mg or 30 mg apremilast twice daily (early escape).
- Apremilast 20 mg: Participants initially randomized to 20 mg apremilast tablets BID in the 24-week placebo-controlled phase, continued receiving 20 mg apremilast tablets twice daily in the active treatment/long-term safety phase. (After 30 mg apremilast BID was identified as the optimal dose, all participants receiving 20 mg apremilast BID were switched to 30 mg apremilast BID dose).
- Apremilast 30 mg: Participants initially randomized to 30 mg apremilast tablets twice daily in the 24-week placebo-controlled phase, continued receiving 30 mg apremilast tablets twice daily in the active treatment / long-term safety phase.
- Placebo / Apremilast 20 mg EE: Participants initially randomized to placebo twice daily in the 24-week placebo-controlled phase were re-randomized due to early escape (EE) at Week 16 and began receiving 20 mg apremilast tablets twice a day in the active treatment phase.
- Placebo / Apremilast 20 mg XO: Participants initially randomized to receive placebo twice daily in the 24-week placebo-controlled phase were re-randomized at Week 24 (XO) to 20 mg apremilast tablets twice daily in the active treatment phase.
- Placebo / Apremilast 30 mg EE: Participants initially randomized to placebo twice daily in the 24-week placebo controlled phase were re-randomized due to early escape (EE) at Week 16 to 30 mg apremilast tablets twice daily in the active-treatment phase.
- Placebo / Apremilast 30 mg XO: Participants initially randomized to placebo twice daily in the 24-week placebo-controlled phase were re-randomized at Week 24 to 30 mg apremilast tablets twice daily in the active treatment phase.
- Placebo/Apremilast 20 mg (Long-Term Safety Phase): Participants initially randomized to placebo tablets twice daily during the placebo controlled phase were re-randomized to 20 mg apremilast twice daily at Week 16 or Week 24 and continued receiving apremilast 20 mg twice daily in the active treatment / long-term safety phase. (After 30 mg apremilast twice daily was identified as the optimal dose, all participants receiving 20 mg apremilast twice daily were switched to the 30 mg apremilast twice daily dose).
- Placebo/Apremilast 30 mg (Long-Term Safety Phase): Participants initially randomized to placebo tablets twice daily during the placebo controlled phase were re-randomized to apremilast 30 mg tablets twice daily at Week 16 or Week 24 and continued receiving apremilast 30 mg twice daily in the active treatment / long-term safety phase.
Period: Placebo-controlled Phase (Week 0 - 24)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 162 | 163 | 163 | 0 | 0 | 0 | 0 | 0 | 0
Received Treatment | 159 | 163 | 162 | 0 | 0 | 0 | 0 | 0 | 0
Completed Week 16 | 148 | 151 | 149 | 0 | 0 | 0 | 0 | 0 | 0
Early Escape at Week 16 | 88 (Two participants who escaped early did not complete Week 24) | 59 (Three participants who escaped early did not complete Week 24) | 64 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 143 (Two participants who completed Week 24 did not enter the active treatment phase) | 143 | 142 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 19 | 20 | 21 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 5 | 12 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomization Error | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Active Treatment Phase (Weeks 24 - 52)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 137 (6 participants who completed Week 24 did not enter the Week 24-52 active treatment phase) | 134 (8 participants who completed Week 24 did not enter the Week 24-52 active treatment phase) | 43 | 27 | 41 (2 participants who EE and completed Week 24 did not enter the Week 24-52 active treatment phase) | 28 | 0 | 0
Completed | 0 | 125 | 114 | 35 | 25 | 34 | 28 | 0 | 0
Not Completed | 0 | 12 | 20 | 8 | 2 | 7 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 3 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 5 | 7 | 4 | 0 | 2 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 7 | 3 | 1 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Long-Term Safety Phase (Year 2)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 119 (6 participants who completed Week 52 did not enter the long-term safety phase) | 109 (5 participants who completed Week 52 did not enter the long-term safety phase) | 0 | 0 | 0 | 0 | 58 (Combined PBO-APR 20EE+XO;2 participants who completed Week 52 did not enter long-term safety phase) | 60 (Combined PBO-APR 30EE+XO;2 participants who completed Week 52 did not enter long-term safety phase)
Completed | 0 | 107 | 95 | 0 | 0 | 0 | 0 | 48 | 51
Not Completed | 0 | 12 | 14 | 0 | 0 | 0 | 0 | 10 | 9
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Lack of Efficacy | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 7 | 9 | 0 | 0 | 0 | 0 | 4 | 6
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Long-Term Safety Phase (Year 3)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 107 | 95 | 0 | 0 | 0 | 0 | 48 | 51
Completed | 0 | 89 | 84 | 0 | 0 | 0 | 0 | 42 | 46
Not Completed | 0 | 18 | 11 | 0 | 0 | 0 | 0 | 6 | 5
Not completed — Adverse Event | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 8 | 5 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2
Period: Long-Term Safety Phase (Year 4)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 89 | 84 | 0 | 0 | 0 | 0 | 41 (1 participant who completed Year 3 did not continue treatment in Year 4) | 46
Completed | 0 | 80 | 77 | 0 | 0 | 0 | 0 | 37 | 39
Not Completed | 0 | 9 | 7 | 0 | 0 | 0 | 0 | 4 | 7
Not completed — Miscellaneous | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Long-Term Safety Phase (Year 5)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo / Apremilast 20 mg EE | Placebo / Apremilast 20 mg XO | Placebo / Apremilast 30 mg EE | Placebo / Apremilast 30 mg XO | Placebo/Apremilast 20 mg (Long-Term Safety Phase) | Placebo/Apremilast 30 mg (Long-Term Safety Phase)
Started | 0 | 80 | 77 | 0 | 0 | 0 | 0 | 38 (1 participant was only counted in year 5 but not in 4 year due to late APR dispensing) | 39
Completed | 0 | 72 | 69 | 0 | 0 | 0 | 0 | 33 | 37
Not Completed | 0 | 8 | 8 | 0 | 0 | 0 | 0 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Non-compliance with study drug | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set consisting of all participants who were randomized as specified in the protocol. Four participants who were randomized in error and did not receive any dose of investigational product are excluded.
Groups:
- Placebo: Participants initially randomized to placebo tablets twice daily in the 24-week placebo-controlled phase. Participants who did not have at least 20% improvement in swollen and tender joint counts at Week 16 were re-randomized to either 20 mg or 30 mg apremilast twice daily (early escape).
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Total
Number analyzed (Participants) | 159 | 163 | 162 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (10.97) | 50.9 (11.82) | 50.5 (11.20) | 50.9 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 95 | 95 | 275
  Male | 74 | 68 | 67 | 209
Duration of Psoriatic Arthritis [Mean (Standard Deviation); unit: years] | 7.76 (8.254) | 7.83 (8.621) | 6.82 (7.592) | 7.47 (8.163)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 16
Description: Percentage of participants with an ACR20 response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 78 tender joint count; • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: Full analysis set consisting of all participants randomized as specified in the protocol; participants who were randomized in error and did not receive any dose of study drug were excluded. Participants who withdrew early or who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
percentage of participants | 18.9 | 37.4 | 32.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; In order to maintain the Type 1 error at the 0.05 significance level, the Hochberg procedure was to be used. The results of the endpoint were to be considered statistically significant if both the 30 mg apremilast dose versus placebo comparison and the 20 mg versus placebo comparison were statistically significant at the 0.05 significance level, or one of the comparisons was statistically significant at the 0.025 level; Test type: Superiority or Other; p = 0.0060, Cochran-Mantel-Haenszel; 2-sided p-value is based on the Cochran-Mantel-Haenszel (CMH) test adjusting for baseline disease modifying antirheumatic drug (DMARD) use; Adjusted Difference = 13.4, 95% CI 2-sided [4.0 to 22.7] — Adjusted difference is the weighted average of the treatment differences across the 2 strata of baseline DMARD use with the CMH weights. The 2-sided 95% confidence interval (CI) is based on a normal approximation to the weighted average
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 18.7, 95% CI 2-sided [9.1 to 28.2] — Adjusted difference is the weighted average of the treatment differences across the 2 strata of baseline DMARD use with the CMH weights. The 2-sided 95% CI is based on a normal approximation to the weighted average

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) at Week 16
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included; Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 153 | 159 | 154
units on a scale | -0.053 (0.0358) | -0.157 (0.0351) | -0.193 (0.0354)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Pairwise comparisons (30 mg vs placebo and 20 mg vs placebo) were conducted conditional on the primary endpoint results. If the primary endpoint was statistically significant for both apremilast dose groups, pairwise comparisons for the HAQ-DI were to be evaluated at the 0.05 level using the Hochberg procedure. If only one apremilast dose was statistically significant, then only the comparison between that apremilast dose and placebo was conducted for the HAQ-DI score, at the 0.025 level; Test type: Superiority or Other; p = 0.0042, ANCOVA; Based on an analysis of covariance (ANCOVA) model with treatment group and baseline DMARD use as factors, and the baseline value as a covariate; LS Mean Difference = -0.140, 95% CI 2-sided [-0.236 to -0.045]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0320, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.104, 95% CI 2-sided [-0.199 to -0.009]

3. Secondary Outcome: Percentage of Participants With an ACR 20 Response at Week 24
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 78 tender joint count; • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦C-Reactive Protein.
Time Frame: Baseline and Week 24
Population: Full analysis set; Participants who discontinued early, escaped early at Week 16 or who did not have sufficient data for a definitive determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
percentage of participants | 15.7 | 31.3 | 24.7
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0394, Cochran-Mantel-Haenszel — Secondary endpoints from the placebo-controlled period (Weeks 16 and 24) were analyzed in a hierarchical fashion to control the Type I error rate as described above; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 9.2, 95% CI 2-sided [0.5 to 17.8] — Adjusted difference is the weighted average of the treatment differences across the 2 strata of baseline DMARD use with the Cochran-Mantel-Haenszel (CMH) weights. The 2-sided 95% CI is based on a normal approximation to the weighted average
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 15.7, 95% CI 2-sided [6.7 to 24.7] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) at Week 24
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 24 are included; LOCF imputation was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 153 | 159 | 154
units on a scale | -0.085 (0.0377) | -0.165 (0.0370) | -0.206 (0.0372)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Secondary endpoints from the placebo-controlled period (Weeks 16 and 24) were analyzed in a hierarchical fashion to control the Type I error rate as described above; Test type: Superiority or Other; p = 0.0191, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.121, 95% CI 2-sided [-0.222 to -0.020]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1179, ANCOVA; LS Mean Difference = -0.080, 95% CI 2-sided [-0.180 to 0.020] — Based on an analysis of covariance (ANCOVA) model with treatment group and baseline DMARD use as factors, and the baseline value as a covariate

5. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) Physical Functioning Domain at Week 16
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 153 | 159 | 153
units on a scale | 0.81 (0.678) | 2.17 (0.664) | 2.91 (0.671)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0237, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 2.10, 95% CI 2-sided [0.28 to 3.92]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1388, ANCOVA; LS Mean Difference = 1.36, 95% CI 2-sided [-0.44 to 3.15] — [estimate comment as in outcome 4, analysis 2]

6. Secondary Outcome: Percentage of Participants With a Modified Psoriatic Arthritis Response Criteria (PsARC) Response at Week 16
Description: Modified PsARC response is defined as improvement in at least 2 of the 4 measures, at least one of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: - 78 tender joint count, - 76 swollen joint count, - Patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest; - Physician global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest. Improvement or worsening in joint counts is defined as decrease or increase, respectively, from baseline by ≥ 30%, and improvement or worsening in global assessments is defined as decrease or increase, respectively, from baseline by ≥ 20 mm VAS.
Time Frame: Baseline and Week 16
Population: Full analysis set; Participants who discontinued early, or who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
percentage of participants | 33.3 | 47.9 | 48.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0065, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 14.9, 95% CI 2-sided [4.3 to 25.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0071, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 14.7, 95% CI 2-sided [4.1 to 25.2] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 16
Description: The participant was asked to place a vertical line on a 100-mm visual analog scale on which the left-hand boundary (score = 0 mm) represents "no pain," and the right-hand boundary (score = 100 mm) represents "pain as severe as can be imagined." The distance from the mark to the left-hand boundary was recorded in millimeters.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 151 | 157 | 152
mm | -7.0 (1.93) | -12.5 (1.89) | -11.9 (1.90)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0648, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -4.9, 95% CI 2-sided [-10.0 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0347, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -5.5, 95% CI 2-sided [-10.6 to -0.4]

8. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 16
Description: The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and at least 1 postbaseline value at or prior to Week 16 are included; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 100 | 105 | 97
units on a scale | -1.0 (0.29) | -0.9 (0.28) | -1.4 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.3496, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.2 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.8874, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.7 to 0.8]

9. Secondary Outcome: Change From Baseline in Dactylitis Severity Score at Week 16
Description: Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet will be rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 16
Population: Full analysis set. Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and at least 1 postbaseline value at or prior to Week 16 are included. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 63 | 75 | 70
units on a scale | -1.1 (0.28) | -0.8 (0.26) | -1.3 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.5438, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-1.0 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.3759, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.3, 95% CI 2-sided [-0.4 to 1.0]

10. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 16
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: - 28 tender joint count (TJC), - 28 swollen joint count (SJC), - Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; - Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8 Low Disease Activity: > 2.8 and ≤ 10 Moderate Disease Activity: > 10 and ≤ 22 High Disease Activity: > 22.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value at or prior to Week 16 are included. LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 149 | 155 | 146
units on a scale | -3.30 (0.871) | -7.75 (0.851) | -6.81 (0.869)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0035, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -3.51, 95% CI 2-sided [-5.86 to -1.16]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0002, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -4.45, 95% CI 2-sided [-6.76 to -2.14]

11. Secondary Outcome: Change From Baseline in the Disease Activity Score (DAS28) at Week 16
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables: - 28 tender joint count - 28 swollen joint count, which do not include the distal interphalangeal (DIP) joints, the hip joint, or the joints below the knee; - C-reactive protein (CRP) - Patient's global assessment of disease activity. DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 16
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 150 | 156 | 151
units on a scale | -0.27 (0.082) | -0.74 (0.080) | -0.67 (0.080)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0004, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.40, 95% CI 2-sided [-0.61 to -0.18]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.47, 95% CI 2-sided [-0.68 to -0.25]

12. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 16
Description: The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue. A positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 153 | 157 | 154
units on a scale | 0.63 (0.724) | 0.91 (0.712) | 2.75 (0.715)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0318, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 2.12, 95% CI 2-sided [0.19 to 4.06]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.7803, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.27, 95% CI 2-sided [-1.65 to 2.20]

13. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) Physical Functioning Domain at Week 24
Description: as for outcome 5
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 153 | 159 | 154
units on a scale | 1.44 (0.688) | 2.97 (0.673) | 3.30 (0.679)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.0473, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 1.86, 95% CI 2-sided [0.02 to 3.70]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.0997, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 1.53, 95% CI 2-sided [-0.29 to 3.35]

14. Secondary Outcome: Percentage of Participants With a Modified Psoriatic Arthritis Response Criteria (PsARC) Response at Week 24
Description: Modified PsARC response is defined as improvement in at least 2 of the 4 measures, at least one of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: • 78 tender joint count, • 76 swollen joint count, • Patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest; • Physician global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest. Improvement or worsening in joint counts is defined as decrease or increase, respectively, from baseline by ≥ 30%, and improvement or worsening in global assessments is defined as decrease or increase, respectively, from baseline by ≥ 20 mm VAS.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
percentage of participants | 24.5 | 39.9 | 32.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.1195, Cochran-Mantel-Haenszel — The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 7.8, 95% CI 2-sided [-1.9 to 17.5] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0026, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 15.5, 95% CI 2-sided [5.6 to 25.5] — [estimate comment as in outcome 1, analysis 2]

15. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 24
Description: as for outcome 7
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 152 | 158 | 153
mm | -8.0 (1.90) | -11.5 (1.86) | -9.7 (1.88)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.5067, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -1.7, 95% CI 2-sided [-6.8 to 3.4]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority or Other; p = 0.1762, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS mean Difference = -3.5, 95% CI 2-sided [-8.5 to 1.6]

16. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 24
Description: as for outcome 8
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and at least 1 postbaseline value at or prior to Week 24 are included; LOCF imputation was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 100 | 105 | 98
units on a scale | -0.9 (0.29) | -0.9 (0.28) | -1.3 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.2719, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-1.2 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.9727, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.0, 95% CI 2-sided [-0.8 to 0.7]

17. Secondary Outcome: Change From Baseline in Dactylitis Severity Score at Week 24
Description: as for outcome 9
Time Frame: Baseline and Week 24
Population: Full analysis set. Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and at least 1 postbaseline value at or prior to Week 24 are included. LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 63 | 75 | 71
units on a scale | -1.1 (0.27) | -0.9 (0.25) | -1.4 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.3705, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.6777, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.6 to 0.8]

18. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 24
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: • 28 tender joint count (TJC), • 28 swollen joint count (SJC), • Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; • Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8; Low Disease Activity: > 2.8 and ≤ 10; Moderate Disease Activity: > 10 and ≤ 22; High Disease Activity: > 22.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 149 | 155 | 148
units on a scale | -3.21 (0.884) | -7.71 (0.864) | -6.35 (0.878)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0097, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -3.14, 95% CI 2-sided [-5.52 to -0.76]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0002, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -4.50, 95% CI 2-sided [-6.85 to -2.16]

19. Secondary Outcome: Change From Baseline in the Disease Activity Score (DAS28) at Week 24
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables: • 28 tender joint count • 28 swollen joint count, which do not include the DIP joints, the hip joint, or the joints below the knee; • C-reactive protein (CRP) • Patient's global assessment of disease activity. DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 150 | 157 | 152
units on a scale | -0.27 (0.084) | -0.73 (0.082) | -0.65 (0.083)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0011, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.38, 95% CI 2-sided [-0.60 to -0.15]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -0.45, 95% CI 2-sided [-0.68 to -0.23]

20. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 153 | 157 | 154
units on a scale | 0.52 (0.721) | 0.68 (0.710) | 2.65 (0.713)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0303, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 2.14, 95% CI 2-sided [0.20 to 4.07]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.8704, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS mean Difference = 0.16, 95% CI 2-sided [-1.76 to 2.08]

21. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 16
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 16 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) are included; LOCF was used. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 104 | 107 | 101
percentage of participants | 52.9 | 54.2 | 56.4
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.6022, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 3.6, 95% CI 2-sided [-9.9 to 17.2] — Adjusted difference is the weighted average of the treatment differences across the 2 strata of baseline DMARD use with the CMH weights
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.8462, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 1.3, 95% CI 2-sided [-12.1 to 14.7] — [estimate comment as in outcome 21, analysis 1]

22. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 16
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 16 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) are included; LOCF was used. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 16 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 66 | 77 | 73
percentage of participants | 59.1 | 62.3 | 61.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.7337, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 2.8, 95% CI 2-sided [-13.3 to 18.9] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.6881, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 3.3, 95% CI 2-sided [-12.7 to 19.3] — [estimate comment as in outcome 3, analysis 1]

23. Secondary Outcome: Percentage of Participants With Good or Moderate European League Against Rheumatism (EULAR) Response at Week 16
Description: A EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score less than or equal to 3.2. A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of less than or equal to 5.1 or, • an improvement (decrease) in the DAS28 of more than 1.2 and attainment of a DAS28 score of greater than 3.2.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
percentage of participants | 31.4 | 53.4 | 48.8
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0014, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 17.5, 95% CI 2-sided [7.0 to 27.9] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 22.1, 95% CI 2-sided [11.7 to 32.5] — [estimate comment as in outcome 1, analysis 2]

24. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 24
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 24 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline MASES > 0 are included; LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 104 | 107 | 101
percentage of participants | 51.0 | 57.0 | 57.4
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.3376, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 6.6, 95% CI 2-sided [-6.8 to 20.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.3756, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 6.1, 95% CI 2-sided [-7.2 to 19.4] — [estimate comment as in outcome 1, analysis 2]

25. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 24
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 24 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Baseline and Week 24
Population: Full analysis set; participants with a baseline dactylitis severity score > 0 are included; LOCF was used. The Week 16 value was carried over to Week 24 for participants who escaped early at Week 16. Participants who did not have sufficient data (observed or imputed) for a determination of response status at Week 24 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 66 | 77 | 73
percentage of participants | 62.1 | 68.8 | 68.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.3959, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 6.8, 95% CI 2-sided [-8.7 to 22.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.3941, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 6.8, 95% CI 2-sided [-8.7 to 22.4] — [estimate comment as in outcome 3, analysis 1]

26. Secondary Outcome: Percentage of Participants With Good or Moderate EULAR Response at Week 24
Description: EULAR response reflects an improvement in disease activity and an attainment of a lower degree of disease activity based on the DAS-28 score. A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score less than or equal to 3.2. A Moderate Response is defined as either: • an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 score of less than or equal to 5.1 or, • an improvement (decrease) in the DAS28 of more than 1.2 and attainment of a DAS28 score of greater than 3.2.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
percentage of participants | 21.4 | 41.7 | 33.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0142, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 12.1, 95% CI 2-sided [2.6 to 21.7] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 20.5, 95% CI 2-sided [10.8 to 30.3] — [estimate comment as in outcome 1, analysis 2]

27. Secondary Outcome: Percentage of Participants With a ACR 50 Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 50% improvement in 78 tender joint count; • ≥ 50% improvement in 76 swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: o Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); o Patient's global assessment of disease activity (measured on a 100 mm VAS); o Physician's global assessment of disease activity (measured on a 100 mm VAS); o Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); o C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
percentage of participants | 5.0 | 14.7 | 10.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.0589, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 5.6, 95% CI 2-sided [-0.2 to 11.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0034, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 9.8, 95% CI 2-sided [3.4 to 16.1] — [estimate comment as in outcome 1, analysis 2]

28. Secondary Outcome: Percentage of Participants With an ACR 70 Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 70% improvement in 78 tender joint count; • ≥ 70% improvement in 76 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: o Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); o Patient's global assessment of disease activity (measured on a 100 mm VAS); o Physician's global assessment of disease activity (measured on a 100 mm VAS); o Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); o C-Reactive Protein.
Time Frame: Baseline and Week 16
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
percentage of participants | 0.6 | 3.7 | 1.2
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.5620, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 0.6, 95% CI 2-sided [-1.5 to 2.7] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.0570, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 3.1, 95% CI 2-sided [-0.0 to 6.2] — [estimate comment as in outcome 1, analysis 2]

29. Secondary Outcome: Percentage of Participants With an ACR 50 Response at Week 24
Description: as for outcome 27
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
percentage of participants | 8.8 | 14.1 | 11.7
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.3629, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 3.1, 95% CI 2-sided [-3.5 to 9.6] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.1323, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 5.4, 95% CI 2-sided [-1.5 to 12.3] — [estimate comment as in outcome 1, analysis 2]

30. Secondary Outcome: Percentage of Participants With a ACR 70 Response at Week 24
Description: Percentage of participants with an American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 70% improvement in 78 tender joint count; • ≥ 70% improvement in 76 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦C-Reactive Protein.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
percentage of participants | 3.1 | 5.5 | 2.5
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.7273, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = -0.6, 95% CI 2-sided [-4.3 to 3.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.2929, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 2.4, 95% CI 2-sided [-2.0 to 6.8] — [estimate comment as in outcome 1, analysis 2]

31. Secondary Outcome: Percentage of Participants Achieving a MASES Score of Zero at Week 16
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 16 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Week 16
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 104 | 107 | 101
percentage of participants | 23.1 | 29.0 | 20.8
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.7023, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = -2.2, 95% CI 2-sided [-13.5 to 9.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.3305, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 5.9, 95% CI 2-sided [-5.9 to 17.7] — [estimate comment as in outcome 1, analysis 2]

32. Secondary Outcome: Percentage of Participants Achieving a Dactylitis Score of Zero at Week 16
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 16 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Week 16
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 66 | 77 | 73
percentage of participants | 40.9 | 42.9 | 41.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.9698, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 0.3, 95% CI 2-sided [-16.0 to 16.6] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.8205, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 1.9, 95% CI 2-sided [-14.3 to 18.1] — [estimate comment as in outcome 1, analysis 2]

33. Secondary Outcome: Percentage of Participants Achieving a MASES Score of Zero at Week 24
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 24 weeks of treatment. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses.
Time Frame: Week 24
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 104 | 107 | 101
percentage of participants | 24.0 | 29.9 | 22.8
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.8424, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = -1.2, 95% CI 2-sided [-12.7 to 10.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.3395, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 5.9, 95% CI 2-sided [-6.0 to 17.8] — [estimate comment as in outcome 1, analysis 2]

34. Secondary Outcome: Percentage of Participants Achieving a Dactylitis Score of Zero at Week 24
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 24 weeks of treatment. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present.
Time Frame: Week 24
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 68 | 59 | 68
percentage of participants | 40.9 | 44.2 | 46.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority; p = 0.4811, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 5.9, 95% CI 2-sided [-10.3 to 22.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 20 mg; Test type: Superiority; p = 0.6965, Cochran-Mantel-Haenszel; The 2-sided p-value is based on the CMH test adjusting for baseline DMARD use; Adjusted Difference = 3.3, 95% CI 2-sided [-13.3 to 19.5] — [estimate comment as in outcome 1, analysis 2]

35. Secondary Outcome: Percentage of Participants With a ACR 20 Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 78 tender joint count; • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population consists of all participants who were randomized or re-randomized to apremilast at any time during the study. Only those participants who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo / Apremilast 20 mg: Participants who received placebo twice daily up to Week 16 or Week 24 were re-randomized to 20 mg apremilast tablets twice daily and continued receiving apremilast 20 mg in the active treatment/long-term phase.
- Placebo / Apremilast 30 mg: Participants who received placebo twice daily up to Week 16 or Week 24 were re-randomized to 30 mg apremilast tablets twice daily and continued receiving apremilast 30 mg in the active treatment/long-term phase.
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 60 | 61 | 121 | 116
percentage of participants | 53.3 [40.0 to 66.3] | 47.5 [34.6 to 60.7] | 52.9 [43.6 to 62.0] | 52.6 [43.1 to 61.9]

36. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 52
Description: as for outcome 2
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a Baseline value and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 60 | 63 | 125 | 117
units on a scale | -0.208 (0.4831) | -0.310 (0.5990) | -0.192 (0.5729) | -0.330 (0.5089)

37. Secondary Outcome: Change From Baseline in the SF-36 Physical Functioning Scale Score at Week 52
Description: as for outcome 5
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 60 | 63 | 124 | 115
units on a scale | 4.13 (9.106) | 5.97 (9.612) | 4.05 (8.752) | 4.97 (9.656)

38. Secondary Outcome: Percentage of Participants With a Modified PsARC Response at Week 52
Description: Modified PsARC response is defined as improvement in at least 2 of the 4 measures, at least one of which must be tender joint count or swollen joint count, and no worsening in any of the 4 measures: • 78 tender joint count, • 76 swollen joint count, • Patient global assessment of disease activity, measured on a 100 mm visual Analog scale (VAS), where 0 mm = lowest disease activity and 100 mm = highest; • Physician global assessment of disease activity, measured on a 100 mm VAS, where 0 mm = lowest disease activity and 100 mm = highest. Improvement or worsening in joint counts is defined as decrease or increase, respectively, from baseline by ≥ 30%, and improvement or worsening in global assessments is defined as decrease or increase, respectively, from baseline by ≥ 20 mm VAS. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; only those participants who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 60 | 60 | 123 | 114
percentage of participants | 78.3 [65.8 to 87.9] | 73.3 [60.3 to 83.9] | 72.4 [63.6 to 80.0] | 74.6 [65.6 to 82.3]

39. Secondary Outcome: Change From Baseline in the Patient Assessment of Pain at Week 52
Description: as for outcome 7
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 60 | 62 | 125 | 117
mm | -15.6 (23.77) | -16.0 (24.48) | -13.5 (27.78) | -12.9 (26.54)

40. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Entheses Score (MASES) at Week 52
Description: as for outcome 8
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a baseline value > 0 (i.e., pre-existing enthesopathy) and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 40 | 39 | 80 | 78
units on a scale | -2.5 (4.41) | -2.5 (2.73) | -1.7 (3.12) | -2.1 (2.82)

41. Secondary Outcome: Change From Baseline in the Dactylitis Severity Score at Week 52
Description: as for outcome 9
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; participants with a baseline value > 0 (i.e., pre-existing dactylitis) and a Week 52 value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 27 | 57 | 60
units on a scale | -1.9 (1.14) | -2.1 (2.32) | -1.8 (1.98) | -1.8 (2.06)

42. Secondary Outcome: Change From Baseline in the CDAI Score at Week 52
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the: • 28 tender joint count (TJC), • 28 swollen joint count (SJC), • Patient's Global Assessment of Disease Activity measured on a 10 cm visual analog scale (VAS), where 0 cm = lowest disease activity and 10 cm = highest; • Physician's Global Assessment of Disease Activity -measured on a 10 cm VAS, where 0 cm = lowest disease activity and 10 cm = highest. The CDAI score ranges from 0-76 where lower scores indicate less disease activity. The following thresholds of disease activity have been defined for the CDAI: Remission: ≤ 2.8 Low Disease Activity: > 2.8 and ≤ 10 Moderate Disease Activity: > 10 and ≤ 22 High Disease Activity: > 22.
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 60 | 60 | 123 | 114
units on a scale | -13.66 (9.811) | -13.13 (13.148) | -12.03 (10.492) | -14.38 (11.531)

43. Secondary Outcome: Change From Baseline in the DAS28 at Week 52
Description: as for outcome 19
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 60 | 62 | 125 | 117
units on a scale | -1.18 (1.015) | -1.18 (1.366) | -1.11 (1.059) | -1.30 (1.033)

44. Secondary Outcome: Change From Baseline in the FACIT-Fatigue Scale Score at Week 52
Description: as for outcome 12
Time Frame: Baseline and Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 59 | 63 | 123 | 115
units on a scale | 1.97 (8.544) | 4.95 (9.414) | 2.45 (9.481) | 4.38 (9.847)

45. Secondary Outcome: Percentage of Participants With MASES Improvement ≥ 20% at Week 52
Description: Percentage of participants with pre-existing enthesopathy whose MASES improved by ≥ 20% from Baseline after 52 weeks. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; only those participants with a baseline MASES > 0 (i.e., pre-existing enthesopathy) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 40 | 39 | 80 | 78
percentage of participants | 72.5 [56.1 to 85.4] | 79.5 [63.5 to 90.7] | 70.0 [58.7 to 79.7] | 69.2 [57.8 to 79.2]

46. Secondary Outcome: Percentage of Participants With Dactylitis Improvement ≥ 1 Point at Week 52
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improved by ≥ 1 after 52 weeks. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; Participants with a baseline dactylitis severity score > 0 (i.e., pre-existing dactylitis) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 27 | 57 | 60
percentage of participants | 95.7 [78.1 to 99.9] | 88.9 [70.8 to 97.6] | 80.7 [68.1 to 90.0] | 85.0 [73.4 to 92.9]

47. Secondary Outcome: Percentage of Participants Achieving Good or Moderate EULAR Response at Week 52
Description: as for outcome 23
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Number; unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 60 | 62 | 125 | 117
percentage of participants | 70.0 | 64.5 | 68.0 | 67.5

48. Secondary Outcome: Percentage of Participants With an ACR 50 Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 50% (ACR50) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 50% improvement in 78 tender joint count; • ≥ 50% improvement in 76 swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 59 | 62 | 120 | 118
percentage of participants | 30.5 [19.2 to 43.9] | 27.4 [16.9 to 40.2] | 26.7 [19.0 to 35.5] | 18.6 [12.1 to 26.9]

49. Secondary Outcome: Percentage of Participants With an ACR 70 Response at Week 52
Description: Percentage of participants with an American College of Rheumatology 70% (ACR70) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 70% improvement in 78 tender joint count; • ≥ 70% improvement in 76 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Baseline and Week 52
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 59 | 63 | 123 | 118
percentage of participants | 16.9 [8.4 to 29.0] | 14.3 [6.7 to 25.4] | 9.8 [5.1 to 16.4] | 6.8 [3.0 to 12.9]

50. Secondary Outcome: Percentage of Participants Achieving a MASES Score of Zero at Week 52
Description: Percentage of participants with pre-existing enthesopathy whose MASES improves to 0 after 24 weeks. The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right. The MASES, ranging from 0 to 13, is the number of painful entheses out of 13 entheses. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Week 52
Population: The Apremilast Subjects as Randomized/Re-randomized (AAR) Population; only those participants with a baseline value > 0 (i.e., pre-existing enthesopathy) and who had sufficient data for a definitive determination of response status at Week 52 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 40 | 39 | 80 | 78
percentage of participants | 42.5 [27.0 to 59.1] | 41.0 [25.6 to 57.9] | 40.0 [29.2 to 51.6] | 37.2 [26.5 to 48.9]

51. Secondary Outcome: Percentage of Participants Achieving a Dactylitis Score of Zero at Week 52
Description: Percentage of participants with pre-existing dactylitis whose dactylitis severity score improves to zero after 52 weeks. Dactylitis is characterized by swelling of the entire finger or toe. Each digit on the hands and feet was rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present. Two-sided 95% confidence interval is based on the Clopper-Pearson method.
Time Frame: Week 52
Population: as for outcome 46
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Apremilast 20 mg | Placebo / Apremilast 30 mg | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 23 | 27 | 57 | 60
percentage of participants | 78.3 [56.3 to 92.5] | 77.8 [57.7 to 91.4] | 57.9 [44.1 to 70.9] | 65.0 [51.6 to 76.9]

52. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events During the Placebo-Controlled Phase
Description: A treatment emergent adverse event (TEAE) is an AE with a start date on or after the date of the first dose of Investigational Product (IP). The severity of each adverse event (AE) and serious AE (SAE) was assessed by the investigator and graded based on a scale from Mild - mild symptoms to Severe AEs (non-serious or serious). A serious adverse event (SAE) is any AE which:
  * Resulted in death
  * Was life-threatening
  * Required inpatient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * Was a congenital anomaly/birth defect
  * Constituted an important medical event
Time Frame: Week 0 to Week 16 for placebo participants who entered EE at Week 16 and up to Week 24 for all other participants (placebo participants who remained on placebo through week 24 and participants randomized to the APR 20 mg BID or APR 30 mg BID)
Population: Safety population included all participants who were randomized and received at least one dose of IP.
Measure: Number; unit: Participants
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 159 | 163 | 162
Participants
  Any TEAE | 72 | 106 | 96
  Any Drug-Related TEAE | 28 | 53 | 57
  Any Severe TEAE | 5 | 3 | 11
  Any Serious TEAE (SAE) | 3 | 6 | 4
  Any Drug-Related SAE | 0 | 3 | 1
  Any TEAE Leading to Drug Interruption | 11 | 16 | 31
  Any TEAE Leading to Drug Withdrawal | 3 | 5 | 12
  Any TEAE Leading to Death | 0 | 0 | 0

53. Secondary Outcome: Number of Participants With TEAEs During the Apremilast-Exposure Period
Description: as for outcome 52
Time Frame: Week 0 to week 260; overall median duration of exposure to apremilast 20 mg and 30 mg BID was 198 weeks
Population: Apremilast subjects as treated who received at least 1 dose of apremilast at any time during the study at week 0, week 16 or week 24.
Measure: Number; unit: participants
Groups:
- Apremilast 20 mg (Pre-switch): Participants who received apremilast 20 mg BID regardless of when the apremilast exposure started (at week 0, 16 and 24). Only the TEAEs that occurred during apremilast 20 mg BID treatment (before the switch to 30 mg apremilast) were included.
- Apremilast 20 mg/30 mg (Post-switch): Participants who switched from apremilast 20 mg BID to apremilast 30 mg BID. Only the TEAEs that occurred during APR 30 mg BID treatment were included.
- Apremilast 30 mg BID: Participants who received apremilast 30 mg twice daily regardless of when the apremilast-exposure started (at Weeks 0, 16, or 24).
Arm/Group | Apremilast 20 mg (Pre-switch) | Apremilast 20 mg/30 mg (Post-switch) | Apremilast 30 mg BID
Number analyzed (Participants) | 234 | 113 | 234
participants
  Any TEAE | 202 | 53 | 207
  Any Drug-related TEAE | 102 | 5 | 100
  Any Severe TEAE | 35 | 2 | 37
  Any Serious TEAE | 41 | 5 | 41
  Any Serious Drug-related TEAE | 6 | 1 | 6
  Any TEAE Leading to Drug Interruption | 47 | 4 | 65
  Any TEAE Leading to Drug Withdrawal | 24 | 3 | 30
  Any TEAE Leading to Death | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: AEs are reported for the placebo-controlled phase from Week 0 to Week 16 for placebo participants who entered EE at Week 16 and up to Week 24 for all other participants. AEs are reported for the Apremilast Exposure Period from Week 0 to Week 260; overall median exposure to apremilast was 198 weeks
Groups:
- Weeks 0-24: Placebo (Placebo-Controlled Phase): Participants received placebo tablets twice daily during the placebo-controlled phase. Includes data through Week 16 for participants who escaped early, and through Week 24 for all other participants.
- Weeks 0-24: Apremilast 20 mg (Placebo- Controlled Phase): Participants received 20 mg apremilast tablets PO BID during the 24-week placebo-controlled phase.
- Weeks 0-24: Apremilast 30 mg (Placebo- Controlled Phase): Participants received 30 mg apremilast tablets PO BID during the 24-week placebo-controlled phase.
- APR Exposure Period Up to 5 Years: APR 20 mg: Participants who received apremilast 20 mg tablets twice daily regardless of when the apremilast exposure started (at Week 0, 16 or 24). Only the TEAEs that occurred during apremilast 20 mg BID treatment (before the switch to 30 mg apremilast) were included.
- APR Exposure Period Up to 5 Years: APR 20mg/30 mg: Participants who switched from apremilast 20 mg BID to apremilast 30 mg BID. Only the TEAEs that occurred during APR 30 mg BID treatment were included.
- APR Exposure Period Up to 5 Years: APR 30 mg: Participants who received 30 mg apremilast twice daily regardless of when their apremilast-exposure started (at Weeks 0, 16, or 24).
Arm/Group | Weeks 0-24: Placebo (Placebo-Controlled Phase) | Weeks 0-24: Apremilast 20 mg (Placebo- Controlled Phase) | Weeks 0-24: Apremilast 30 mg (Placebo- Controlled Phase) | APR Exposure Period Up to 5 Years: APR 20 mg | APR Exposure Period Up to 5 Years: APR 20mg/30 mg | APR Exposure Period Up to 5 Years: APR 30 mg
Serious Adverse Events (participants affected / at risk) | 3/159 | 6/163 | 4/162 | 41/234 | 5/113 | 41/234
Other Adverse Events (participants affected / at risk) | 38/159 | 73/163 | 82/162 | 154/234 | 19/113 | 166/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weeks 0-24: Placebo (Placebo-Controlled Phase) (N=159) | Weeks 0-24: Apremilast 20 mg (Placebo- Controlled Phase) (N=163) | Weeks 0-24: Apremilast 30 mg (Placebo- Controlled Phase) (N=162) | APR Exposure Period Up to 5 Years: APR 20 mg (N=234) | APR Exposure Period Up to 5 Years: APR 20mg/30 mg (N=113) | APR Exposure Period Up to 5 Years: APR 30 mg (N=234)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abscess soft tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Neuroborreliosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Peritoneal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Scrotal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Skin candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 3
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Brain stem stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Carotid artery disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 3 | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Weeks 0-24: Placebo (Placebo-Controlled Phase) (N=159) | Weeks 0-24: Apremilast 20 mg (Placebo- Controlled Phase) (N=163) | Weeks 0-24: Apremilast 30 mg (Placebo- Controlled Phase) (N=162) | APR Exposure Period Up to 5 Years: APR 20 mg (N=234) | APR Exposure Period Up to 5 Years: APR 20mg/30 mg (N=113) | APR Exposure Period Up to 5 Years: APR 30 mg (N=234)
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 2 | 14 | 0 | 9
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4 | 5 | 11 | 1 | 13
Diarrhoea (Gastrointestinal disorders) | 8 | 18 | 25 | 33 | 0 | 40
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 5 | 12 | 0 | 12
Nausea (Gastrointestinal disorders) | 3 | 15 | 26 | 25 | 1 | 37
Vomiting (Gastrointestinal disorders) | 2 | 5 | 6 | 10 | 1 | 12
Bronchitis (Infections and infestations) | 0 | 5 | 6 | 19 | 1 | 30
Influenza (Infections and infestations) | 0 | 4 | 3 | 13 | 0 | 10
Nasopharyngitis (Infections and infestations) | 6 | 9 | 9 | 28 | 4 | 30
Pharyngitis (Infections and infestations) | 2 | 1 | 2 | 8 | 1 | 15
Rhinitis (Infections and infestations) | 1 | 1 | 1 | 5 | 0 | 13
Sinusitis (Infections and infestations) | 4 | 4 | 3 | 17 | 1 | 15
Upper respiratory tract infection (Infections and infestations) | 6 | 14 | 11 | 42 | 4 | 37
Urinary tract infection (Infections and infestations) | 2 | 3 | 1 | 18 | 4 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 14 | 0 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3 | 22 | 0 | 14
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 11 | 2 | 12
Headache (Nervous system disorders) | 7 | 9 | 18 | 23 | 0 | 29
Depression (Psychiatric disorders) | 2 | 1 | 0 | 13 | 0 | 7
Insomnia (Psychiatric disorders) | 0 | 3 | 1 | 14 | 0 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 3 | 12 | 0 | 15
Hypertension (Vascular disorders) | 7 | 4 | 5 | 21 | 4 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.